CLINICAL TRIAL: NCT04696380
Title: Do Flavors Increase the Addiction Potential of Nicotine?: A Pilot Laboratory Study
Brief Title: Do Flavors Increase the Addiction Potential of Nicotine?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, John Hughes, MD, Professor, University of Vermont
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: CHRMS 00000555
Record Dates: First submitted 2020-11-23; First posted 2021-01-06 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Nicotine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- High nicotine, preferred flavor (Experimental): Participants will sample their preferred flavored JUUL e-cigarette at 5% nicotine strength.
  Interventions: Drug: Nicotine; Device: JUUL e-cigarette
- High nicotine, non-preferred flavor (Experimental): Participants will sample their non-preferred flavored JUUL e-cigarette at 5% nicotine strength.
  Interventions: Drug: Nicotine; Device: JUUL e-cigarette
- Low nicotine, preferred flavor (Experimental): Participants will sample their preferred flavored JUUL e-cigarette at 3% nicotine strength.
  Interventions: Drug: Nicotine; Device: JUUL e-cigarette
- Low nicotine, non-preferred flavor (Experimental): Participants will sample their non-preferred flavored JUUL e-cigarette at 3% nicotine strength.
  Interventions: Drug: Nicotine; Device: JUUL e-cigarette

INTERVENTIONS:
Drug: Nicotine — Participants will sample high vs low nicotine.
Device: JUUL e-cigarette — Participants will sample preferred vs non-preferred JUUL flavors.

SUMMARY:
The FDA has concluded that flavors (e.g. menthol) are associated with greater addiction potential in tobacco cigarettes (Gottlieb March 13, 2019). Whether the same is true for e-cigarettes and non-menthol flavors is unclear and our study should help answer this question.

Our major hypothesis is that the pharmacological effect of nicotine to induce addiction will be greater with use of a preferred e-cigarette flavor than with use of a non-preferred flavor. The pharmacological effect will be measured by how much a larger nicotine dose increases addiction potential compared to a smaller dose.

DETAILED DESCRIPTION:
Study Design:

Fifteen participants who currently use e-cigarettes weekly and who use or do not use tobacco cigarettes will enter a remote session study. Participants will be asked to abstain from all nicotine/tobacco products, non-nicotine electronic cigarettes, and THC containing products for 16 hours prior to four experimental sessions and will be tested in a 2x2 within-participants design with four conditions: 1) low nicotine dose (3%)/non-preferred flavor, 2) low dose/preferred flavor, 3) high dose (5%)/non-preferred flavor, and 4) high dose/preferred flavor. Order of testing will be randomized. Participants and experimenters will be blind to dose. The major outcomes will be subjective effects, e.g. liking and tests of reinforcement (choice procedures). We will require 16 hours of abstinence prior to each remote experimental session to increase the sensitivity to nicotine effects.

The consent process, experimental sessions and data collection will all be done remotely using a secure video platform. The only interaction between participants and research staff will be the curbside pick-up of study products, which will follow social distancing and mask guidelines. Participants will pick up study JUUL pods curb-side at the University of Vermont before their baseline videoconference session. Participants will be required to conduct all videoconference sessions in a place where they can legally use their JUUL.

The consent videoconference session will be conducted prior to the baseline and four experimental sessions. Participants will be assessed for COVID-19 and E-cigarette or Vaping Product Use-Associated Lung Injury (EVALI) symptoms prior to the curbside pick-up and at the start of the 5 videoconference sessions in which they will be asked to vape. During the baseline session, participants will complete a baseline questionnaire via online survey and then answer a series of questions about nicotine dependence and how many JUUL pods they would purchase at varying prices. Participants will then sample the two flavors available for JUUL -Virginia Tobacco and Menthol- using their own JUUL device. Research staff will ask participants to rate the pleasantness of each flavor and, after they have tried the flavors, participants will rank order their flavor preferences to determine their preferred flavor of the two. Finally, participants will be trained in the puffing protocol to be used in the experimental sessions.

During each experimental videoconference session, participants will report on their recent e-cigarette and tobacco product use at the start of each videoconference testing session. Those reporting non-abstinence will have their videoconference session rescheduled. During the videoconference testing sessions participants will be asked to puff either tobacco flavor 3% nicotine, tobacco flavor 5% nicotine, menthol flavor 3% nicotine, or menthol flavor 5% nicotine. After each puffing bout within each session, they will answer questions about about e-cigarette effects, e-cigarette liking and wanting, like/dislike of e-cigarette taste and e-cigarette intensity. At the end of each session, they will be asked how many JUUL pods they would purchase at varying prices.

Adverse events will be collected at the end of each videoconference session by the research assistant, who will consult with the study licensed medical provider.

ELIGIBILITY:
Inclusion criteria:

* 21 years or older
* comfortable reading and writing English
* own a JUUL brand e-cigarette they have used at least 10 times in the past 30 days
* use JUUL e-cigarettes and JUUL pods with 5% nicotine
* used e-cigarettes on 4+ days a week in the last 30 days
* use or do not use tobacco cigarettes
* do not plan to quit e-cigarettes in the next 30 days
* non-pregnant females verified by pregnancy test
* access to the internet in a location where they could join a videoconference call and legally use their JUUL.
* Reside in VT

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Liking and wanting nicotine | 2 weeks
  Average of "I feel good e-cigarette effects", "I want more of that e-cigarette I received", "I feel the e-cigarette strength" and "I like the e-cigarette effect" on a 0-100mm scale from "not at all" (0) to "extremely" (100).
E-cigarette purchase task | 2 weeks
  This is a modification of the Cigarette Purchase Task that asks how much users would spend to obtain their usual amount of e-liquids to use.
E-cigarette and tobacco cigarette craving | 2 weeks
  Modified items from the Mood and Physical Symptoms Scale that asks about change/strength of urges for e-cigarettes and tobacco cigarettes (0-4 scale, 0= not at all and 4= extremely) and strength of urges (1-5 scale, 1=slight and 5= extremely strong).
Modified Drug Effect Questionnaire | 2 weeks
  Modified version of the Drug Effects Questionnaire where participants rate acute responses to the e-cigarette drug effects on a 0-100 mm scale, from "not at all" (0) to "extremely" (100).
Modified Labeled Hedonic Scale | 2 weeks
  1 item about like/dislike of the e-cigarette taste using a modified version of the Labeled Hedonic Scale, a category ratio scale that ranges from -100 (most disliked) to 100 (most liked).
Modified Labeled Magnitude Scale | 2 weeks
  1 item about e-cigarette taste intensity using a modified version of the Labeled Magnitude Scale, which is a category ratio scale with 7 semantic labels: "no sensation", "barely detectable", "weak", "moderate", "strong", "very strong", and "strongest imaginable", with responses coded on a 0-100 scale (0= no sensation, 100= strongest imaginable).

CONTACTS AND LOCATIONS:
Overall Officials: John R Hughes, MD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peasley-Miklus C, Klemperer EM, Hughes JR, Villanti AC, Krishnan-Sarin S, DeSarno MJ, Mosca LA, Su A, Cassidy RN, Feinstein MJP. The interactive effects of JUUL flavor and nicotine concentration on addiction potential. Exp Clin Psychopharmacol. 2023 Apr;31(2):336-342. doi: 10.1037/pha0000591. Epub 2022 Sep 1. PMID 36048114